CLINICAL TRIAL: NCT06182722
Title: Association of Peripheral Immune Cells With Antidepressant Treatment Response
Status: Recruiting | Type: Observational
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, LI, Huafang, Principal Investigator, Shanghai Mental Health Center
Other Study IDs: 2022-TX-010
Record Dates: First submitted 2023-09-16; First posted 2023-12-27 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Depressive Disorder; Genetic Change
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples With DNA — Peripheral blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Major Depressive Disorder (MDD): Patients with major depressive disorder. These patients consisted of two cohorts. The first cohort is expected to consist of 15 participants for nested cohort study. The rest form the second cohort.
  Interventions: Diagnostic Test: Mental assessments
- Healthy controls: Healthy normal volunteers.

INTERVENTIONS:
Diagnostic Test: Mental assessments — Patients will receive psychiatric rating scales evaluation every visit.
  Other Names: Psychiatric rating scales
  Groups: Major Depressive Disorder (MDD)

SUMMARY:
The purpose of this observational study is discovering potential biomarkers to predict antidepressant treatment response in patients with major depressive disorder (MDD) while comparing the transcriptomic changes between patients with MDD and healthy controls as well as before and after antidepressant treatment.

Eligible patients will be assessed at Week 1, Week 2, Week 4 and Week 8 while healthy normal volunteers will only be evaluated at baseline. Assessments will include the following: an interview about mental and physical health, a physical examination including drawing of venous blood samples and several psychiatric rating scales.

DETAILED DESCRIPTION:
This study is focusing on evaluating the peripheral immune system of major depressive disorder (MDD) and the impact of antidepressants treatment. Single-cell RNA sequencing and single-cell VDJ sequencing will be performed on peripheral blood mononuclear cells to collect transcriptome information and immune repertoire of peripheral blood in patients with MDD. Bulk RNA sequencing and flow cytometry will be used to validate the clinical value of results.

This is a biomarker study (antidepressants); treatment will be carried out according to physicians' orders.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old, regardless of gender;
2. The subject is an outpatient/inpatient and meets DSM-5 diagnostic criteria of current or past major depressive disorder;
3. SSRIs or SNRIs monotherapy;
4. HAMD-17 total score ≥ 18 at baseline;
5. The subject can read and write and is capable of giving informed consent.

Exclusion Criteria:

1. Patients with mental illness other than MDD;
2. Patients with liver and kidney diseases, cardiovascular system diseases, cancer, diabetes, thyroid diseases or other serious or unstable conditions;
3. Previous organic brain disease, traumatic brain injury or other diseases that can cause structural brain changes;
4. Serious abnormalities indicated by laboratory tests or electrocardiograms;
5. Alcohol or drug addiction;
6. Suffering from systemic lupus erythematosus, multiple sclerosis or other autoimmune diseases;
7. Patients who are taking drugs that directly impact on the immune system such as anti-inflammatory drugs or immunosuppressants;
8. Patients who have taken antidepressants or other antipsychotics within 2 weeks before enrollment;
9. Patients who have received MECT or systematic psychotherapy within 3 months before enrollment;
10. Patients at high risk of suicide, or reporting a HAMD-17 item 3 (suicide item) score >3 at baseline;
11. Subjects who are pregnant or lactating;
12. Other conditions that are considered not suitable for participating in the research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatients/inpatients who meet DSM-5 diagnostic criteria of current or past major depressive disorder and are going to receive SSRIs or SNRIs monotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change of HAMD-17 (Hamilton Depression Rating Scale) total score | From baseline to Week 8
  The overall score of HAMD-17 (Hamilton Depression Rating Scale) is 68 points. Primary outcome measures the change of HAMD-17 total score between baseline and week 8. Larger reduction in HAMD-17 represents better antidepressant treatment response.

SECONDARY OUTCOMES:
Effective rate measured by HAMD-17 (Hamilton Depression Rating Scale) | From baseline to Week 8
  A reduction of 50% or more in the HAMD-17 (Hamilton Depression Rating Scale) total score. More patients with a reduction of 50% or more indicates better effectiveness. Minimun value of HAMD-17 is 0 and maximum value of HAMD-17 is 68 points.
MADRS Effective rate measured by MADRS (Montgomery-Åsberg depression rating scale) | From baseline to Week 8
  A reduction of 50% or more in the MADRS (Montgomery-Åsberg depression rating scale) total score. More patients with a reduction of 50% or more indicates better effectiveness. Minimun value of MADRS is 0 and maximum value of MADRS is 60 points.
Remission rate measured by HAMD-17 (Hamilton Depression Rating Scale) | From baseline to Week 8
  HAMD-17 (Hamilton Depression Rating Scale) total score ≤10 at week8. Lower total score of HAMD-17 at week 8 indicates better outcome. Minimun value of HAMD-17 is 0 and maximum value of HAMD-17 is 68 points.
MADRS Remission rate measured by MADRS (Montgomery-Åsberg depression rating scale) | From baseline to Week 8
  MADRS (Montgomery-Åsberg depression rating scale) total score ≤7 at week8. Lower total score of HAMD-17 at week 8 indicates better outcome. Minimun value of MADRS is 0 and maximum value of MADRS is 60 points.

OTHER OUTCOMES:
HAMD-17 (Hamilton Depression Rating Scale) total score | Baseline, Week 2, Week 4 and Week 8.
  Minimun value of HAMD-17 (Hamilton Depression Rating Scale) is 0 and maximum value of HAMD-17 is 68 points. Higher scores implies higher severity.
MADRS (Montgomery-Åsberg depression rating scale) total score | Baseline, Week 2, Week 4 and Week 8.
  Minimun value of MADRS (Montgomery-Åsberg depression rating scale) is 0 and maximum value of MADRS is 60 points. Higher scores implies higher severity.
CGI-S (Clinical Gloabl Impression-Severity) score | Baseline, Week 2, Week 4 and Week 8.
  Minimun value of CGI-S (Clinical Gloabl Impression-Severity) is 0 and maximum value of CGI-S is 7 points. Higher scores implies higher severity.
CGI-I (Clinical Gloabl Impression-Improvement) score | Baseline, Week 2, Week 4 and Week 8.
  Minimun value of CGI-I (Clinical Gloabl Impression-Improvement) is 1 points and maximum value of CGI-I is 7 points. Higher scores implies worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Shen He, Study Director — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

REFERENCES:
- [Background] Malhi GS, Mann JJ. Depression. Lancet. 2018 Nov 24;392(10161):2299-2312. doi: 10.1016/S0140-6736(18)31948-2. Epub 2018 Nov 2. PMID 30396512
- [Background] Kato T, Furukawa TA, Mantani A, Kurata K, Kubouchi H, Hirota S, Sato H, Sugishita K, Chino B, Itoh K, Ikeda Y, Shinagawa Y, Kondo M, Okamoto Y, Fujita H, Suga M, Yasumoto S, Tsujino N, Inoue T, Fujise N, Akechi T, Yamada M, Shimodera S, Watanabe N, Inagaki M, Miki K, Ogawa Y, Takeshima N, Hayasaka Y, Tajika A, Shinohara K, Yonemoto N, Tanaka S, Zhou Q, Guyatt GH; SUN☺D Investigators. Optimising first- and second-line treatment strategies for untreated major depressive disorder - the SUN☺D study: a pragmatic, multi-centre, assessor-blinded randomised controlled trial. BMC Med. 2018 Jul 11;16(1):103. doi: 10.1186/s12916-018-1096-5. PMID 29991347
- [Background] Leday GGR, Vertes PE, Richardson S, Greene JR, Regan T, Khan S, Henderson R, Freeman TC, Pariante CM, Harrison NA; MRC Immunopsychiatry Consortium; Perry VH, Drevets WC, Wittenberg GM, Bullmore ET. Replicable and Coupled Changes in Innate and Adaptive Immune Gene Expression in Two Case-Control Studies of Blood Microarrays in Major Depressive Disorder. Biol Psychiatry. 2018 Jan 1;83(1):70-80. doi: 10.1016/j.biopsych.2017.01.021. Epub 2017 Jul 6. PMID 28688579
- [Background] Nohr AK, Lindow M, Forsingdal A, Demharter S, Nielsen T, Buller R, Moltke I, Vitezic M, Albrechtsen A. A large-scale genome-wide gene expression analysis in peripheral blood identifies very few differentially expressed genes related to antidepressant treatment and response in patients with major depressive disorder. Neuropsychopharmacology. 2021 Jun;46(7):1324-1332. doi: 10.1038/s41386-021-01002-9. Epub 2021 Apr 8. PMID 33833401
- [Background] Cattaneo A, Ferrari C, Turner L, Mariani N, Enache D, Hastings C, Kose M, Lombardo G, McLaughlin AP, Nettis MA, Nikkheslat N, Sforzini L, Worrell C, Zajkowska Z, Cattane N, Lopizzo N, Mazzelli M, Pointon L, Cowen PJ, Cavanagh J, Harrison NA, de Boer P, Jones D, Drevets WC, Mondelli V, Bullmore ET; Neuroimmunology of Mood Disorders and Alzheimer's Disease (NIMA) Consortium; Pariante CM. Whole-blood expression of inflammasome- and glucocorticoid-related mRNAs correctly separates treatment-resistant depressed patients from drug-free and responsive patients in the BIODEP study. Transl Psychiatry. 2020 Jul 23;10(1):232. doi: 10.1038/s41398-020-00874-7. PMID 32699209
- [Background] Zheng C, Zheng L, Yoo JK, Guo H, Zhang Y, Guo X, Kang B, Hu R, Huang JY, Zhang Q, Liu Z, Dong M, Hu X, Ouyang W, Peng J, Zhang Z. Landscape of Infiltrating T Cells in Liver Cancer Revealed by Single-Cell Sequencing. Cell. 2017 Jun 15;169(7):1342-1356.e16. doi: 10.1016/j.cell.2017.05.035. PMID 28622514